CLINICAL TRIAL: NCT02787967
Title: A Single-dose, Open-label, Randomized, 2-way Cross-over Study of CHF 1535 35/4 NEXThaler® (Fixed Combination of Beclometasone Dipropionate (BDP) 35 μg Plus Formoterol Fumarate (FF) 4 μg Versus the Free Combination of Licensed BDP DPI (Dry Powder Inhaler) and FF DPI in Asthmatic Children
Brief Title: Clinical Pharmacology of 35/4 NEXThaler® in Children 5-11 Years Old
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CCD-01535BB1-01; 2015-005152-10 (EudraCT Number)
Record Dates: First submitted 2016-03-15; First posted 2016-06-02 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NEXThaler® 35/4µg (Experimental): CHF 1535 35/4µg NEXThaler® Dry Powder Inhaler, 4 inhalations. Total Dose: BDP 200µg FF 16µg
  Interventions: Drug: CHF 1535 35/4µg NEXThaler®
- Reference treatment (Active Comparator): Drug: free comb. beclomethasone DPI and formoterol DPI 2 (two) inhalations BDP 100 µg DPI + 4 (four) inhalations FF 6 µg DPI (total dose: BDP 200 µg + FF 24 µg
  Interventions: Drug: free comb. beclomethasone DPI and formoterol DPI

INTERVENTIONS:
Drug: CHF 1535 35/4µg NEXThaler® — 4 (four) inhalations (total dose: BDP/FF 140/16 µg)
  Arms: NEXThaler® 35/4µg
Drug: free comb. beclomethasone DPI and formoterol DPI — 2 (two) inhalations BDP 100 µg DPI + 4 (four) inhalations FF 6 µg DPI (total dose: BDP 200 µg + FF 24 µg
  Arms: Reference treatment

SUMMARY:
The study will be conducted in asthmatic children aged 5 to 11 years and is based on a single-dose, open-label, randomized, 2-way cross-over design where a Dry Powder Inhaler (DPI) fixed combination of beclometasone dipropionate (BDP) 35 μg plus formoterol fumarate (FF) 4 μg is compared with the free combination of licensed BDP DPI and FF DPI

DETAILED DESCRIPTION:
This is a pharmacokinetic comparison of NEXThaler 35/4 μg versus the free combination of Beclomethasone DPI and Formoterol DPI in children (5 to 11 years old) of a formulation already approved in adults.

ELIGIBILITY:
Inclusion Criteria:

* Male/female children with asthma stable enough, according to paediatrician opinion, to allow a wash out period from steroids of 3 days before study treatments.
* Male/female children with asthma on regular treatment with ICS or using short-acting inhaled 2-agonist as reliever to control asthma symptoms.
* Age ≥ 5 < 12 years (8 to 10 children in the age range 5-8 years old).
* Children with a forced expiratory volume in one second (FEV1)>70% of predicted values (% pred) after withholding 2-agonists treatment for a minimum of 4 h prior to screening and to each study treatment.
* A cooperative attitude and ability to be trained about the proper use of DPI, ability to use correctly the medical devices and compliant to study procedures

Exclusion Criteria:

* Past or present diagnosis of cardiovascular, renal or liver disease.
* Known hypersensitivity to the active treatmen
* Exacerbation of asthma symptoms within 4 weeks prior to screening.
* Inability to perform the required breathing technique and blood sampling.
* Hospitalization due to exacerbation of asthma within 1 month prior to screening (Visit 1).
* Lower respiratory tract infection within 1 month prior to screening (Visit 1).
* Disease (other than asthma) which might influence the outcome of the study.
* Obesity, i.e. > 97% weight percentile by local standards

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2016-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Plasma Area Under Curve (AUC0-t) for B17MP, active metabolite of BDP | predose, 15,30min, 1,2,4,6,8 hours post dose
  B17MP: Profile of Pharmacokinetics

SECONDARY OUTCOMES:
B17MP Cmax | predose, 15min,30min,1,2,4,6,8 hours post dose
  17MP: profile of pharmacokinetics
BDP Area Under Curve (AUC) | predose, 15min,30min,1,2,4,6,8 hours post dose
  BDP: profile of Pharmacokinetics
Formoterol Area Under Curve (AUC), Cmax, Tmax, T1/2 [ | predose, 15min, 30 min, 1,2,4,6,8 hours postdose
  Formoterol: profile of pharmacokinetics
Formoterol Cmax | predose, 15min, 30 min, 1,2,4,6,8 hours postdose
  Formoterol: profile of pharmacokinetics
Formoterol Tmax | predose, 15min, 30 min, 1,2,4,6,8 hours postdose
  Formoterol: profile of pharmacokinetics
Formoterol T1/2 | predose, 15min, 30 min, 1,2,4,6,8 hours postdose
  Formoterol: profile of pharmacokinetics
plasma potassium Area Under Curve (AUC) | predose, 15min, 30min, 1, 2, 4, 6, 8 hours postdose
  plasma potassium to evaluate drug systemic effect
plasma potassium Cmin | predose, 15min, 30min, 1, 2, 4, 6, 8 hours postdose
  plasma potassium to evaluate drug systemic effect
plasma potassium Tmin | predose, 15min, 30min, 1, 2, 4, 6, 8 hours postdose
  plasma potassium to evaluate drug systemic effect
Urinary Cortisol: Amount excreted in 0-8hours (Ae),8h cortisol urinary excretion normalized for 8h creatinine excretion (Ae/Aecreat). | from predose up to 8 hours postdose
  Urinary cortisol to evaluate drug systemic effect
B17MP Tmax | predose, 15min,30min,1,2,4,6,8 hours post dose
  BDP: profile of pharmacokinetics
B17MP T1/2 | predose, 15min,30min,1,2,4,6,8 hours post dose
  BDP: profile of pharmacokinetics
BDP Cmax | predose, 15min,30min,1,2,4,6,8 hours post dose
  BDP: profile of pharmacokinetics
BDP Tmax | predose, 15min,30min,1,2,4,6,8 hours post dose
  BDP: profile of pharmacokinetics
BDP T1/2 | predose, 15min,30min,1,2,4,6,8 hours post dose
  BDP: profile of pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Hans Bisgaard, MD, Principal Investigator — Copenhagen Studies on Asthma in Childhood
Locations (1):
- BørneAstmaKlinikken, Hans Knudsens Plads 1A,, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2015-005152-10/results